CLINICAL TRIAL: NCT00417976
Title: A Phase II Study of the Combination of Fixed Dose Rate Gemcitabine, Infusional 5 Fluorouracil and Bevacizumab in Patients With Advanced Pancreas Cancer
Brief Title: Gemcitabine, Infusional 5 Fluorouracil and Bevacizumab in Patients With Advanced Pancreas Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tony Bekaii-Saab (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Tony Bekaii-Saab, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-05110; NCI-2011-03230 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Results first posted 2014-11-03 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Pancreatic Cancer
Keywords: Advanced Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Bevacizumab; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Experimental)
  Interventions: Drug: Gemcitabine; Drug: Bevacizumab; Drug: Infusional 5-Fluorouracil

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m2 over 100 minutes every 2 weeks.
  Other Names: Gemzar
Drug: Bevacizumab — 10 mg/kg every 2 weeks.
  Other Names: Avastin
Drug: Infusional 5-Fluorouracil — 2400 mg/m2 over 48 hours every 2 weeks.
  Other Names: Adrucil; Efudex; Fluoroplex

SUMMARY:
This is a phase II study of biweekly (every other week) bevacizumab followed by gemcitabine then infusional 5-fluorouracil in patients with stage III or IV pancreatic cancer. Patients' response will be evaluated every 8 weeks using usual CT scanning techniques. RECIST (Response Evaluation Criteria in Solid tumors) criteria will be applied to evaluate response. Tumor marker levels (Ca 19-9) will be assessed every 4 weeks, but will not be used to measure response.

DETAILED DESCRIPTION:
Rationale: Research indicates that the vascular endothelial growth factor (VEGF), or a substance made by cells that stimulates new blood vessel formation, plays an important role in the growth and metastasis of many cancers, including pancreatic carcinoma. Both VEGF and its receptors are overexpressed in pancreatic cancer. Bevacizumab works by blocking VEGF and the growth of cancer cells in the process. The current study combines bevacizumab with two commonly used pancreatic cancer drugs, gemcitabine and infusional 5-FU. Previous studies indicate that bevacizumab combined with other anti-cancer drugs such as 5-FU improves patient survival. In addition, other research suggests that the drug administration schedule of the current study may improve patient outcomes compared to other types of administration and sequencing.

Purpose: The primary objective of this study is to assess the rate of progression free survival at 6 months in patients with advanced pancreatic cancer given gemcitabine, infusional 5-FU, and bevacizumab. Secondary objectives of this study include measuring response rates, 6 month and 1-year survival rates, and median overall survival.

Treatment: Study participants will be given bevacizumab, gemcitabine, and 5-FU. These drugs will be administered through intravenous infusions in that order every other week on days 1 and 15. Treatments will be given in 28-day cycles. Participants will therefore receive study drugs during weeks 1 and 3, and then receive no study drugs during weeks 2 and 4. Imaging exams will be performed every 8 weeks to assess disease size. Several other tests will be given throughout the study to closely monitor patients. Tumor level markers will be assessed every 4 weeks, but will not be used to measure response. Study treatments will be discontinued due to disease growth or severe adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age >=18 years.
* Established histological confirmation of adenocarcinoma of the pancreas.
* Stage III and stage IV will be allowed.

Exclusion Criteria:

* No prior chemotherapy or radiotherapy allowed except for that given as part of an adjuvant regimen if >4 weeks have elapsed since the end of therapy. Any prior treatment with antibodies to VEGF.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to starting the study.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-12; Primary Completion 2010-03 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanios Saab, M.D., Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The University of Michigan, Ann Arbor, Michigan
  - The Ohio State University James Cancer Hospital, Columbus, Ohio

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab: Gemcitabine : 1000 mg/m2 over 100 minutes every 2 weeks.
  Bevacizumab : 10 mg/kg every 2 weeks.
  Infusional 5-Fluorouracil : 2400 mg/m2 over 48 hours every 2 weeks.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 42
Completed | 39
Not Completed | 3
Not completed — Non compliance unrelated to toxicity | 1
Not completed — Treatment -related toxicity | 2

BASELINE CHARACTERISTICS:
Population: 42 patients enrolled in study; of which, 39 were evaluable for primary end point.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 60 [36 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 40
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 42
Eastern Cooperative Oncology Group (ECOG) Performance status [Number; unit: participants]
  0 (Fully Active) | 15
  1 (Restricted in physical activity) | 27
Site of metastasis [Number; unit: participants]
  Liver only | 29
  Liver+other | 2
  Other only | 9
  Recurrent metastatic disease | 2
Prior adjuvant therapy [Number; unit: participants]
  Gemcitabine-based | 1
  Chemoraditation | 1
  No prior adjuvant therapy | 40
Disease stage [Number; unit: participants]
  III (Unresectable primary tumor) | 2
  IV (Cancer has spread o distant tissue or organ) | 40
CA19-9 (tumor marker levels) [Number; unit: participants]
  Normal (≤37 U/ml) | 6
  Elevated (>37 U/ml) | 36
Albumin [Number; unit: participants]
  Normal (≥3.4 g/dl) | 28
  Low (<3.4 g/dl) | 14

OUTCOME MEASURES:

1. Primary Outcome: Rate of Progression Free Survival at 6 Months (24 Weeks) From Initiation of Therapy
Time Frame: 6 months
Measure: Number; unit: percent of patients
Arm/Group | Bevacizumab
Number analyzed (Participants) | 39
percent of patients | 49

2. Secondary Outcome: Response Rates Defined by RECIST 1.0
Description: The National Cancer Institutes Response Evaluation Criteria in Solid Tumors (RECIST) 1.0 was used in accessing response for patients
Time Frame: 6 months
Measure: Number; unit: patients
Arm/Group | Bevacizumab
Number analyzed (Participants) | 40
patients
  Complete Respsonse | 0
  Partial Response | 12
  Stable Disease | 18
  Progressive Disease | 10

ADVERSE EVENTS:
Time Frame: Adverse events were graded according to the NCI-CTCAE (Common Toxicity Criteria for Adverse Effects) v 3.0. Toxicity assessments were repeated on day 1 and 15 of every cycle.
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 1/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=42)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=42)
Anemia (Blood and lymphatic system disorders) | 27 (27)
Thrombocytopenia (Injury, poisoning and procedural complications) | 13 (13)
Leukopenia (Investigations) | 11 (11)
Neutropenia (Investigations) | 6 (6)
Lymphopenia (Investigations) | 8 (8)
Fatigue (General disorders) | 26 (26)
Vomiting (Gastrointestinal disorders) | 33 (33)
Nausea (Gastrointestinal disorders) | 25 (25)
Diarrhea (Gastrointestinal disorders) | 16 (16)
Elevated ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 7 (7)
Elevated AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 6 (6)
Mucositis (Gastrointestinal disorders) | 9 (9)
Altered sense of taste (Nervous system disorders) | 12 (12)
Hypertension (Vascular disorders) | 8 (8)
Fistula formation (Gastrointestinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Bleeding (Vascular disorders) | 7 (7)
Thrombosis (Vascular disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
42 patients enrolled, 39 were evaluable for the primary end point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No